CLINICAL TRIAL: NCT04573387
Title: A Randomized Controlled Trial of Exhaustive Drainage Versus Fixed-time Drainage for Chronic Subdural Hematoma After One-burr Hole Craniostomy
Brief Title: Exhaustive Drainage Versus Fixed-time Drainage for Chronic Subdural Hematoma After One-burr Hole Craniostomy
Acronym: ECHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Weiming Liu, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY 2020-094-02
Record Dates: First submitted 2020-09-26; First posted 2020-10-05 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Hematoma, Subdural, Chronic
Keywords: chronic subdural hematoma; fixed-time drainage; exhaustive drainage; drainage; craniostomy; urokinase
MeSH Terms: conditions — Hematoma, Subdural, Chronic | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The design is open labeled with only the investigators for postoperative follow-up evaluation, the outcome assessors, and data analysts being blinded in all 19 centers. Before outcome assessment begins at every follow-up evaluation, the patients will be reminded not to reveal any information about their group allocation. If details of group allocation can be detected by the investigator during follow-ups, another blinded researcher will replace to evaluate outcome.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fixed-time drainage (Active Comparator): Drainage will be removed after 48 hours.
  Interventions: Procedure: Operation; Procedure: Fixed-time drainage; Procedure: Postoperative computed tomography
- Exhaustive drainage (Experimental): Drainage will be removed when postoperative hematoma volume is minimized with repeated urokinase injection into hematoma cavity through catheter.
  Interventions: Procedure: Operation; Procedure: Exhaustive drainage; Procedure: Postoperative computed tomography

INTERVENTIONS:
Procedure: Operation — All participants are treated with burr-hole craniotomy and a drainage system as follows. Participants undergo surgical procedure under local anesthesia in the hemisphere with a lateral position, but general anesthesia is performed when participant cannot tolerate the operation. A single 1.5 cm burr hole is drilled over the maximum width of the hematoma cavity. After coagulating with bipolar diathermy, dura mater is opened with a cruciate incision. A soft catheter is placed carefully in all directions of the hematoma cavity for irrigating subdural collections with 1,000 mL warm Ringer's lactate saline until clarification. The drainage catheter is inserted ½ length of the maximum diameter of the hematoma cavity toward the frontal region. After the skin is closed, the catheter was connected to a soft collection bag that is placed under the head for passive drainage. During the drainage period, participants stay in bed until the drain is removed.
Procedure: Fixed-time drainage — All participants will be treated with a one-burr-hole craniotomy with irrigation and a closed drainage system. The drainage will be removed after 48 hours.
  Arms: Fixed-time drainage
Procedure: Exhaustive drainage — All participants will be treated with a one-burr-hole craniotomy with irrigation and a closed drainage system. If the computed tomography (CT) scan on the first day after surgery indicates that the affected brain region shows sufficient re-expansion, the drainage catheter will be removed when drainage ceases. If subdural collections remain in the hematoma cavity, the participant will be treated with 30,000 U urokinase injection into the hematoma cavity through the catheter. The catheter will be closed and reopened in 1.5-2 hours, and a CT scan will be performed when drainage ceases. If the CT scan shows sufficient re-expansion of the brain, the catheter will be removed. However, if the brain does not show good re-expansion and there is still a residual subdural collection, the above steps will be repeated. If the participant is subjected to urokinase injection for 3 times, the catheter will be removed when drainage ceases.
  Arms: Exhaustive drainage
Procedure: Postoperative computed tomography — All participants undergo a CT scan before the drain is removed, and the last CT scan will be performed before the patient is discharged from the hospital.

SUMMARY:
A prospective, multicenter, randomized controlled trial is designed to compare the recurrence rates and clinical outcomes in patients with chronic subdural hematoma using exhaustive drainage or fixed-time drainage after one-burr hole craniostomy.

DETAILED DESCRIPTION:
Chronic subdural hematomas (CSDHs) are one of the most common neurosurgical conditions. The goal of surgery is to alleviate symptoms and minimize the risk of symptomatic recurrences. The standard surgical technique includes burr-hole craniostomy, followed by intraoperative irrigation and placement of subdural closed-system drainage. The drainage is removed after 48 hours, which can be described as fixed-time drainage strategy. According to literature, the recurrence rate is 5-33% with this strategy. In the investigators' retrospective study, postoperative hematoma volume (p=0.001, B=0.028, Exp(B)=1.028, 95% CI 1.011-1.046) was found to significantly increase the risk of recurrence. Based on these results, an exhaustive drainage strategy may minimize postoperative hematoma volume and achieve a low recurrence rate and good outcomes. This is a prospective, multicenter, randomized controlled trial designed to include 304 participants over the age of 18 years presenting with a symptomatic CSDH verified on cranial computed tomography or magnetic resonance imaging. After informed consent is obtained, participants are randomly allocated to an exhaustive drainage or fixed-time drainage group. The primary endpoint is recurrence indicating a reoperation within 6 months. Secondary outcomes include modified Rankin Scale, Markwalder Grading Scale, European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L), rate of complications, rate of adverse events and effect on comorbidity.

ELIGIBILITY:
Inclusion Criteria:

* Patient (18 years to 90 years) presenting with clinical symptoms and neurological deficits of chronic subdural hematoma
* Chronic subdural hematoma verified on cranial computed tomography or magnetic resonance imaging
* Written informed consent from patients or their next of kin according to the patient's cognitive status

Exclusion Criteria:

* No clinical symptoms correlating with chronic subdural hematoma
* Lack of mass effect, less than 0.5 cm of midline structure shift, and no need surgery judged clinically by neurosurgeons
* Previous surgery for chronic subdural hematoma during the past 6 months
* Previous intracranial surgery for any neurological disorders but chronic subdural hematoma before
* Existing poor medication condition or severe comorbidity so that surgery cannot be tolerated or follow-up cannot be completed
* Severe coagulopathy or high risk of life-threatening bleeding
* Postoperative cooperation is suspected to be insufficient for follow-up for 6 months
* Reproductive-age women without verified negative pregnancy testing
* Participating in other research

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Rate of re-operations of chronic subdural hematoma | From operation up to 6 months postoperatively
  Rate of re-operations between fixed-time drainage group and exhaustive drainage group

SECONDARY OUTCOMES:
Change of Modified Rankin Scale (MRS) between groups from baseline to 6 months after operation | At baseline, and at 1, 3, and 6 months after operation
  Modified Rankin Scale ranges from score 1 to 6, and higher scores mean a worse clinical outcome, where score 1 indicates normal daily functionality and score 6 indicates death.
Change of Markwalder Grading Scale (MGS) between groups from baseline to 6 months after operation | At baseline, and at 1, 3, and 6 months after operation
  Markwalder Grading Scale ranges from grade 0 to 4, and higher scores mean a worse neurological outcome, where grade 0 indicates normal neurological function and grade 4 indicates coma.
Change of health related quality of life between groups from baseline to 6 months after operation | At baseline, and at 1, 3, and 6 months after operation
  A standardized instrument, EuroQoL 5-Dimension 5-Level (EQ-5D-5L) questionnaire, will be used as a generic measure of health related quality of life. The questionnaire contains 5 dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Each dimension rates across five levels, including 'No problems-Slight problems-Moderate problems-Severe problems-Unable to'.
Rate of mortality between groups within 6 months | From operation up to 6 months postoperatively
  Rate of mortality between fixed-time drainage group and exhaustive drainage group
Rate of complications and adverse events between groups within 6 months | From operation up to 6 months postoperatively
  Rate of complications and adverse events between fixed-time drainage group and exhaustive drainage group within 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Weiming Liu, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (17):
- China (17):
  - Beijing Ditan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Luhe Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Wangjing Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - Puning People's Hospital, Puning, Guangdong
  - Wei County Hospital of Traditional Chinese Medicine, Handan, Hebei
  - Hengshui People's Hospital, Hengshui, Hebei
  - First Hospital of Qinhuangdao, Qinhuangdao, Hebei
  - North China University of Science and Technology Affiliated Hospital, Tangshan, Hebei
  - Xiahuayuan District Hospital, Zhangjiakou, Hebei
  - First People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - Yancheng Third People's Hospital, Yancheng, Jiangsu
  - People's Hospital of Ningxia Hui Autonomous Region, Yinchuan, Ningxia
  - Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ou Y, Yu X, Liu X, Jing Q, Liu B, Liu W. A Comparative Study of Chronic Subdural Hematoma in Patients With and Without Head Trauma: A Retrospective Cross Sectional Study. Front Neurol. 2020 Nov 27;11:588242. doi: 10.3389/fneur.2020.588242. eCollection 2020. PMID 33329333
- [Background] Ou Y, Dong J, Wu L, Xu L, Wang L, Liu B, Li J, Liu W. An Exhaustive Drainage Strategy in Burr-hole Craniostomy for Chronic Subdural Hematoma. World Neurosurg. 2019 Jun;126:e1412-e1420. doi: 10.1016/j.wneu.2019.03.111. Epub 2019 Mar 19. PMID 30902781
- [Background] Ou Y, Dong J, Wu L, Xu L, Wang L, Liu B, Li J, Liu W. The Clinical Characteristics, Treatment, and Outcomes of Chronic Subdural Hematoma in Young Patients. World Neurosurg. 2019 May;125:e1241-e1246. doi: 10.1016/j.wneu.2019.02.017. Epub 2019 Feb 22. PMID 30797913
- [Background] Ou Y, Dong J, Wu L, Xu L, Wang L, Liu B, Li J, Liu W. A comparative study of chronic subdural hematoma in three age ranges: Below 40 years, 41-79 years, and 80 years and older. Clin Neurol Neurosurg. 2019 Mar;178:63-69. doi: 10.1016/j.clineuro.2019.01.018. Epub 2019 Jan 29. PMID 30716602
- [Background] Liu W, Bakker NA, Groen RJ. Chronic subdural hematoma: a systematic review and meta-analysis of surgical procedures. J Neurosurg. 2014 Sep;121(3):665-73. doi: 10.3171/2014.5.JNS132715. Epub 2014 Jul 4. PMID 24995782
- [Background] Wu L, Ou Y, Liu W. Letter to the Editor. Benefit of postoperative computed tomography in chronic subdural hematoma. J Neurosurg. 2019 Sep 13;131(6):1992-1993. doi: 10.3171/2019.5.JNS191212. Print 2019 Dec 1. No abstract available. PMID 31518980
- [Derived] Wu L, Ou Y, Zhu B, Guo X, Yu X, Xu L, Li J, Feng E, Li H, Wang X, Chen H, Sun Z, Liu Z, Yang D, Zhang H, Liu Z, Tang J, Zhao S, Zhang G, Yao J, Ma D, Sun Z, Zhou H, Liu B, Liu W; ECHO Trial Collaborators. Exhaustive drainage versus fixed-time drainage for chronic subdural hematoma after one-burr hole craniostomy (ECHO): study protocol for a multicenter randomized controlled trial. Trials. 2023 Mar 20;24(1):207. doi: 10.1186/s13063-023-07250-y. PMID 36941714